CLINICAL TRIAL: NCT04995900
Title: Heart Matters: A Stepped-wedge Cluster Randomized Controlled Trial of Heart Health Education Targeting Communities at High Risk of Acute Coronary Syndrome.
Brief Title: Heart Matters: The Effectiveness of Heart Health Education in Regions at Highest-risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Heart Foundation, Australia (Other); Department of Health, Victorian Government (Unknown); Ambulance Victoria (Other Government)
Responsible Party: Principal Investigator, Janet, Associate Professor, Monash University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 291276657; 1180282 (Other Grant/Funding Number: National Health and Medical Research Council (NHMRC))
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction, Acute
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: The stepped-wedge design is a uni-directional cross-over design - where the randomisation element is when the cluster crosses-over to the intervention following a control period.
Who Masked: Outcomes Assessor
Masking Description: Outcomes are collected blinded to the study allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention period with active Heart Matters education delivered
  Interventions: Other: Community education
- Control (No Intervention): Control period with no Heart Matters education delivered.

INTERVENTIONS:
Other: Community education — Heart Matters coordinators will deliver heart health education to the community using HM materials and Partner resources.
  Other Names: Local campaign
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate whether providing a targeted heart health education campaign to regions at high risk of heart attacks will improve ACS patient's symptom recognition and response.

The intervention will be will be evaluated according to a cluster randomized, stepped wedged design. The clusters are eight local government areas (LGAs) in Victoria, Australia. The main primary outcome will be assessed in consecutive patients presenting to emergency departments from the six LGAs throughout the study period with an ED diagnoses of acute coronary syndrome.

DETAILED DESCRIPTION:
Primary objectives:

To determine if targeted heart health education will:

1. Increase ambulance use in ACS patients (main primary outcome);
2. Decrease patient and prehospital delay times in ACS patients;
3. Increase awareness of personal cardiovascular risk and associated factors in adult community members; and
4. Increase cardiovascular knowledge and confidence to act to heart attack warning signs in adult community members.

Secondary objectives

1. To determine if targeted heart health education:
2. Reduces the incidence of out-of-hospital cardiac arrest;
3. Improves survival in OHCA patients;
4. Improves survival in ACS patients;
5. Improves survival and ACS patients;
6. Increases presentations to ED for ACS and unspecified chest pain; and
7. Increases the rates of calls to ambulance for chest pain and non-chest pain.
8. Increases the rate of Heart Health Checks.

Intervention: To meet the objectives of the study, we will employ HM coordinators for each of the eight high-risk LGAs to organise and deliver our HM education program using HM materials and Partner resources.

Design: The stepped-wedge design is a uni-directional cross-over design - where the randomisation element is when the cluster crosses-over to the intervention following a control period.

Over the 16-month study period, the eight LGAs will move into the intervention phase at two month intervals. As four LGAs are in close proximity, these LGAs will switch from control to intervention periods at the same time to avoid possible contamination.

ELIGIBILITY:
Inclusion Criteria: Adult residents of the eight local government areas -

Exclusion Criteria: Adults not residing in the eight local government areas.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2240 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Ambulance use for ACS | 16 months
  The proportion of ACS patients that present to ED by ambulance.

SECONDARY OUTCOMES:
Median ACS patient delay time | 16 months
  The median ACS patients delay time (time from symptom onset to decision to seek medical attention).
ACS patient delay time <60 minutes | 16 months
  The proportion of ACS patients with patient delay times <60 minutes
Median ACS patient prehospital delay time | 16 months
  The median ACS patient prehospital delay time (time from symptom onset to arrival at hospital).
ACS patients prehospital delay times <120 minutes | 16 months
  The proportion of ACS patients with prehospital delay times <120 minutes
Awareness of own risk of heart attack | 0-2 months and 6-8 months
  The proportion of adult members of the community who are aware of their own risk of heart attack.
Awareness of heart attack as a leading cause of death | 0-2 months and 6-8 months
  The proportion of adult members of the community who identify heart disease a leading cause of death
Awareness of heart attack risk factors | 0-2 months and 6-8 months
  The proportion of adult members of the community who identify cardiovascular risk factors
Number of correctly named heart attack risk factors | 0-2 months and 6-8 months
  The number of correctly named cardiovascular risk factors by adult members of the community
Awareness of heart attack signs and symptoms | 0-2 months and 6-8 months
  The proportion of adult members of the community aware of heart attack symptoms
Number of correctly named heart attack signs and symptoms | 0-2 months and 6-8 months
  The number of correctly named ACS symptoms by adult members of the community
Confidence in knowing how to act | 0-2 months and 6-8 months
  The proportion adult members of the community who are confident about what they would do if experiencing a heart attack
Ambulance use in scenarios | 0-2 months and 6-8 months
  The proportion adult members of the community who correctly state they would call an ambulance for two heart attack scenarios.
Rates of Heart Health Checks | 16 months
  Rates of Medicare claims for General Practitioner (GP) Heart Health Checks
Rates of ACS ED presentations | 16 months
  The rates of ED presentations that are ACS
Rates of unspecified chest pain ED presentations | 16 months
  Rates of ED presentations that are unspecified chest pain
ACS ED presentations via GPs | 16 months
  Proportion of ACS ED presentations via General Practitioners
Rates of ACS survival | 16 months
  The proportion of ACS patients surviving to hospital discharge
Incidence of OHCA | 16 months
  incidence of out-of-hospital cardiac arrest
Rates of OHCA | 16 months
  Rates out-of-hospital cardiac arrest survival
Calls to ambulance for chest pain | 16 months
  Proportion of chest pain (event type 10) calls to ambulance
Calls to ambulance for non- chest pain | 16 months
  Proportion of non-chest pain emergency calls to ambulance

CONTACTS AND LOCATIONS:
Locations (1):
- Victorian LGAs, Melbourne, Please Select, Australia

IPD SHARING:
Plan to Share IPD: No
Access to data is restricted and is not available for sharing at the individual patient level.

REFERENCES:
- [Derived] Bray JE, Nehme Z, Finn JC, Kasza J, Clark RA, Stub D, Cadilhac DA, Buttery AK, Woods J, Kim J, Smith BJ, Smith K, Cartledge S, Beauchamp A, Dodge N, Walker T, Flemming-Judge E, Chow C, Stewart M, Cox N, van Gaal W, Nadurata V, Cameron P. A protocol for the Heart Matters stepped wedge cluster randomised trial: The effectiveness of heart attack education in regions at highest-risk. Resusc Plus. 2023 Jul 25;15:100431. doi: 10.1016/j.resplu.2023.100431. eCollection 2023 Sep. PMID 37555197